CLINICAL TRIAL: NCT05172791
Title: Decreasing Unnecessary Antibiotics Prescribed for Possible Pneumonia Despite Normal Respiratory Rate and Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Klompas, M.D., Medical Doctor, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2021p002282
Record Dates: First submitted 2021-12-01; First posted 2021-12-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2023-08

CONDITIONS: Pneumonia
Keywords: antibiotic stewardship; pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual care (No Intervention): Clinical teams will decide on antibiotic duration for patients with possible pneumonia without external prompting
- Electronic alert (Experimental): An electronic alert will be displayed within the electronic medical record of eligible patients that notes that the patient's respiratory rate and oxygenation are within the normal range and will advise stopping antibiotics prescribed for possible pneumonia
  Interventions: Behavioral: Antibiotic stewardship messaging
- Pharmacist (Experimental): Pharmacists will contact the treating teams of eligible patients to note that the patient's respiratory rate and oxygenation are within the normal range and will advise stopping antibiotics prescribed for possible pneumonia.
  Interventions: Behavioral: Antibiotic stewardship messaging

INTERVENTIONS:
Behavioral: Antibiotic stewardship messaging — Counseling regarding antibiotics for patients prescribed antibiotics for possible pneumonia despite respiratory rates and oxygenation levels within normal ranges
  Arms: Electronic alert; Pharmacist

SUMMARY:
The purpose of this study is to decrease unnecessary antibiotics prescribed to hospitalized patients for possible pneumonia by flagging patients with respiratory rates and oxygenation levels within reference ranges given prior data suggesting that discontinuing antibiotics in this population is safe. Patients will be randomized to 3 arms: 1) usual care, 2) electronic alert, or 3) pharmacist outreach.

DETAILED DESCRIPTION:
Prior data suggest antibiotic starts for patients with normal vital signs are common and there does not appear to be harm associated with stopping antibiotics after only 1 or 2 days in patients with normal oxygen saturations. We therefore propose a pilot patient-level three-way randomized trial to determine the best way to operationalize professional society recommendations for post-prescription antibiotic reviews amongst patients started on antibiotics with a stated indication of pneumonia despite normal respiratory rates and oxygenation levels. If the patient's median respiratory rate and oxygen saturation is normal after 1-2 days of antibiotics they will be randomized to usual care versus a EHR-based best practice alert versus pharmacist outreach. The EHR-based best practice alert will highlight the patient's normal respiratory rate and oxygenation and encourage stopping antibiotics if there isn't another indication for antibiotics. Pharmacist outreach will involve contacting the responding clinician or attending physician to determine the working diagnosis, review the patient's vital signs, and to ask the team to consider stopping antibiotics if there are no clear indications for antibiotics. In all cases, the final decision on whether to stop or continue antibiotics will be up to the primary team. We will assess the impact of these post-prescription review strategies to decrease unnecessary antibiotic utilization on antibiotic utilization (antibiotic days and antibiotic-free days) compared to usual care. Safety outcomes will include time to discharge, readmissions, hospital-free days, and mortality. We will also assess for change in the primary outcome over time.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Brigham and Women's and BWH Faulkner Hospitals and prescribed antibiotics with a stated indication of pneumonia who have a median respiratory rate of ≤20 and oxygen saturation of ≥95% without supplemental oxygen sustained for at least 24 hours.

Exclusion Criteria:

* Patients under 18 years old, patients on transplant and oncology services, patients who are pregnant, patients in an intensive care unit, patients with cystic fibrosis or bronchiectasis, patients on immunosuppressive medications, and patients with positive blood cultures (other than common skin contaminants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Duration of antibiotics prescribed for pneumonia | Number of days of antibiotics given during hospitalization plus number of days of antibiotics for pneumonia on discharge prescriptions, up to 30 days
  Duration of antibiotics prescribed for pneumonia

SECONDARY OUTCOMES:
Antibiotic-free days in the 30-days post-randomization | 30-days post-randomization
  Antibiotic-free days in the 30-days post-randomization
Days from randomization to discharge | Duration of hospitalization, up to 90 days
  Days from randomization to discharge
Hospital length of stay | Duration of hospitalization, up to 90 days
  Hospital length of stay
In-hospital mortality | During initial hospitalization with pneumonia, up to 90 days
  In-hospital mortality
Readmissions within 30-days of randomization | 30-days post-randomization
  Readmissions within 30-days of randomization
Hospital-free days in the 30-days post-randomization | 30-days post-randomization
  Hospital-free days in the 30-days post-randomization
C. difficile infections in the 30-days post-randomization | 30-days post-randomization
  C. difficile infections in the 30-days post-randomization
Acute kidney injury (maximum creatinine in the 14-days post-randomization) | 14 days post-randomization
  Acute kidney injury (maximum creatinine in the 14-days post-randomization)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Klompas, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No